CLINICAL TRIAL: NCT04776759
Title: Atrial Fibrillation in Young Patients: a Prospective Multicentre Registry
Acronym: YOUNG-AF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Rythmo20200901
Record Dates: First submitted 2020-09-03; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-08

CONDITIONS: Atrial Fibrillation; Lone Atrial Fibrillation
Keywords: Atrial Fibrillation; Lone Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation is a rare cardiac arrhythmia in young (i.e. <= 35-year-old) patients. Etiological factors, current management and mid- to long-term outcomes remain unknown.

DETAILED DESCRIPTION:
Atrial Fibrillation in YOUNG patients (YOUNG-AF) is a prospective, observational, multicentric registry, including every consecutive patients aged < 35-year-old with a diagnosis of atrial fibrillation. The registry will assess demographical, physical activity, toxicologic and genetic factors, as well as current management regarding anticoagulation, anti-arrhythmic drugs and catheter ablation. As an observational registry, patient will be managed with the guidelines-directed standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* First episode of atrial fibrillation
* Less than 35-year-old
* Diagnostic by 12-lead ECG or continuous monitoring (minimal duration 30 seconds)
* French Social Security number

Exclusion Criteria:

* Transvenous cardiac implantable electronic device (insertable cardiac monitors are not an exclusion criteria)

Max Age: 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Young patients (i.e. < or = to 35-year-old) at the time of first atrial fibrillation episode.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite of mortality, thromboembolic event and heart failure | at 10-year
  Incidence of all-cause mortality, symptomatic thromboembolic event and congestive heart failure at 10-year after initial diagnosis of atrial fibrillation.
Recurrent symptomatic atrial fibrillation. | at 10-year
  Incidence of symptomatic atrial fibrillation at 10-year after initial diagnosis of atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No